CLINICAL TRIAL: NCT03144375
Title: Comparison of Outcomes After Peri-operative Optimization and Standard Surgical Treatment or Standard of Care Surgical Treatment in Patients Who Have Chronic Rhinosinusitis With Polyposis.
Brief Title: QOL Outcomes in CRS With Polyps
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: inability to promptly see local allergists as part of medical maximization which lead to delays in care for these patients
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Corinna Levine, Assistant Professor, University of Miami
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 20151068
Record Dates: First submitted 2017-05-03; First posted 2017-05-08 (Actual); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Chronic Rhinosinusitis, Polyps
MeSH Terms: conditions — Polyps | interventions — Educational Status

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Medical Optimization (Active Comparator): Medical treatment and education x 4 months, re- eval at 4 months and possible cross-over to surgery
  Interventions: Other: Medical optimization and education; Procedure: Standard of Care sinus surgery
- Surgical treatment (Active Comparator): Surgical treatment up front
  Interventions: Procedure: Standard of Care sinus surgery

INTERVENTIONS:
Other: Medical optimization and education — Medical treatment and education about the sinusitis disease process prior to surgery as compared to baseline surgical and treatment counseling
  Arms: Medical Optimization
Procedure: Standard of Care sinus surgery

SUMMARY:
Chronic rhinosinusits (CRS) is common disease with reports of prevalence ranging from 4-16% in the western population. The main outcome measure for chronic disease treatment, such as CRS, is quality of life. Several large multi-institutional studies have shown that improvement in disease specific Quality of life was greater in patients who had surgery for their CRS with polyps. The timing of surgery in these patients has not been well studied but it is generally agreed upon that surgical candidates much had failed medical management. The definition of medical management varies greatly but usually includes some form of nasal or oral steroids and a prolonged ( >10 days) course of antibiotics.

Another known way to improve QOL is through education and individualized optimization. This has been utilized successfully in other fields with good success and improved QOL. Similar studies looking at combining non-surgical optimization and education have not been performed in CRS. This study aims to address this potential area for improvement in patient quality of life outcomes. Investigators plan to assess the potential role for pre-operative non-surgical medical and educational optimization in CRS standard of care treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adults with Rhinosinusitis with polyps who have had appropriate treatment qualifying them for surgery and are good surgical candidates

Exclusion Criteria:

* Cystic fibrosis, Cilia disorders, other specialized forms of sinus disease

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-12; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
SNOT-22 | 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Miami, Miami, Florida, United States